CLINICAL TRIAL: NCT05018806
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multicenter Proof-of-concept Study Evaluating Efficacy and Safety of Rilzabrutinib in Adult Patients With Moderate-to-severe Atopic Dermatitis Who Are Inadequate Responders or Intolerant to Topical Corticosteroids
Brief Title: Proof of Concept Study of Rilzabrutinib in Adult Patients With Moderate-to-severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT17207; U1111-1261-7565 (Registry Identifier: ICTRP); ACT17207 (Other: Sanofi Identifier); 2021-001704-15 (EudraCT Number)
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BID cohort: Placebo (Placebo Comparator): Participants received placebo matched to rilzabrutinib orally BID from Day 1 up to Week 16. Consecutive doses were ideally administered 12 hours apart (and not less than 8 hours apart).
  Interventions: Drug: Placebo
- BID cohort: Rilzabrutinib (Experimental): Participants received rilzabrutinib 400 milligrams (mg) orally BID from Day 1 up to Week 16. Consecutive doses were ideally administered 12 hours apart (and not less than 8 hours apart).
  Interventions: Drug: Rilzabrutinib
- TID cohort: Placebo (Placebo Comparator): Participants received placebo matched to rilzabrutinib orally TID from Day 1 up to Week 16. Consecutive doses were ideally administered at least 6 hours apart (and not less than 4 hours apart).
  Interventions: Drug: Placebo
- TID cohort: Rilzabrutinib (Experimental): Participants received rilzabrutinib 400 mg orally TID from Day 1 up to Week 16. Consecutive doses were ideally administered at least 6 hours apart (and not less than 4 hours apart).
  Interventions: Drug: Rilzabrutinib

INTERVENTIONS:
Drug: Placebo — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: BID cohort: Placebo; TID cohort: Placebo
Drug: Rilzabrutinib — Pharmaceutical form: Tablet Route of administration: Oral
  Other Names: PRN1008/SAR444671
  Arms: BID cohort: Rilzabrutinib; TID cohort: Rilzabrutinib

SUMMARY:
This was a parallel treatment, Phase 2, double-blind, 2-arm, placebo-controlled study with 2 staggered cohorts (2 arms in each cohort) to evaluate the efficacy and safety of rilzabrutinib in adult participants (aged at least 18 years) with moderate-to-severe AD and intolerance or inadequate response to topical corticosteroids (TCS).

The total study duration per participant was expected to be approximately 21 weeks, including up to 4 weeks of screening, 16 weeks of on-treatment double-blind period, 1 week of post-treatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

* AD as defined by the American Academy of Dermatology Consensus Criteria.
* History of AD for at least 12 months prior to baseline as determined by the Investigator through patient interview.
* Eczema Area and Severity Index (EASI) score ≥ 12 at screening and at baseline.
* IGA score ≥ 3 (on the 0 to 4 IGA scale) at baseline.
* BSA of AD involvement ≥ 10% at baseline.
* Documented inadequate response or intolerance to TCS within 6 months prior to baseline visit
* Baseline PP-NRS score for maximum itch intensity ≥4.
* All contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* For optional substudy only: Willingness to have 2 tape strips for comparison of baseline and treatment response.

Exclusion Criteria:

* Skin comorbidities that may interfere with study assessments such as psoriasis, tinea corporis, lupus erythematosus.
* Conditions that may predispose the patient to excessive bleeding.
* Any other clinically significant disease, condition, or medical history that, in the opinion of the Investigator, would interfere with participant safety, trial evaluations, and/or trial procedures.
* Laboratory abnormalities at the screening visit
* History of serious infections requiring intravenous therapy with the potential for recurrence (as judged by the Site Investigator and the Sponsor Medical Monitor), with less than 4 weeks interval between resolution of serious infection and first dose of study drug, or currently active moderate to severe infection at Screening (Grade 2 or higher) including active coronavirus disease 2019 (COVID-19).
* Live vaccine except Bacille Calmette Guerin-vaccination within 28 days prior to Day 1 or plan to receive one during the trial; Bacille Calmette Guerin-vaccination within 12 months prior to Screening.
* COVID-19 vaccine within 14 days prior to Study Day 1.
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate rilzabrutinib/placebo absorption.
* Initiation of prescription moisturizers (with or without additives such as ceramide, hyaluronic acid, urea, or filaggrin), topical anesthetics or antihistamines during the screening period.
* Use of TCS, topical calcineurin (tacrolimus, and/or pimecrolimus) or topical phosphodiesterase 4 inhibitor within 1 week prior to baseline and as concomitant medication.
* Use of systemic corticosteroids within 4 weeks prior to baseline and as concomitant medication.
* Phototherapy for AD or regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks prior to baseline or likely to be required as concomitant procedure during the study.
* Use of mycophenolate mofetil, azathioprine, methotrexate, cyclosporine, dapsone, intravenous immunoglobulin (IVIG), Kineret (anakinra), Enbrel (etanercept), or any other immunosuppressant not mentioned in this exclusion criterion within 4 weeks prior to baseline.
* Use of infliximab, adalimumab, golimumab, abatacept, tocilizumab, certolizumab, secukinumab, IFN-γ, JAK inhibitors, dupilumab, and any other biologic or targeted-synthetic disease modifier drug not mentioned in this exclusion criterion or in exclusion criterion, as well as plasmapheresis within 12 weeks prior to baseline.
* Use of anti-CD20 drugs such as rituximab, ofatumumab, other long-acting biologics within 6 months prior to baseline (or shorter if there is documented B cell reconstitution for anti-CD20 drugs).
* Use of proton pump inhibitor drugs such as omeprazole and esomeprazole within 3 days of baseline (it is acceptable to change participant to H2 receptor blocking drugs prior to baseline).
* Concomitant use of known systemic strong-to-moderate inhibitors and inducers of cytochrome P450 3A (CYP3A) within 14 days or 5 half-lives (whichever is longer) prior to baseline.
* Previous use of a BTK inhibitor.
* Had received any investigational drug (or is currently using an investigational device) within the 30 days before baseline, or at least 5 times the respective elimination half-life time (whichever is longer).
* Active TB or a history of incompletely treated TB, Quantiferon positive patients, Clinically significant abnormality consistent with prior/active TB infection based upon chest radiograph with at least posterior-anterior view, Suspected extrapulmonary TB infection, or patients at high risk of contracting TB.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline to Week 16 in Eczema Area and Severity Index (EASI) Score | Baseline (Day 1) to Week 16
  The EASI index is a validated investigator-administered scoring system used to measure the severity of clinical signs in atopic dermatitis (AD). Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) were each assessed for severity by the investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement were assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. 0: 0% of body surface area (BSA) involvement with AD; 1: 1-9%; 2: 10-29%; 2: 30-49%; 4: 50-69%; 5: 70-89% and 6: 90-100% of BSA involvement with AD. Total score ranged from 0 (minimum) to 72 (maximum); higher scores indicated greater severity of AD. Baseline was defined as the Day 1 assessment value.

SECONDARY OUTCOMES:
Percentage of Participants With Investigator's Global Assessment (IGA) of 0 or 1 At Week 16 | Week 16
  IGA is a static 5-point measure of disease severity based on an overall assessment of the skin lesions on a 5-point scale (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). Higher score indicated higher severity.
Percentage of Participants Achieving EASI-75 (Reduction of EASI Score By ≥75% From Baseline) At Week 16 | Baseline (Day 1) and at Week 16
  The EASI index is a validated investigator-administered scoring system used to measure the severity of clinical signs in AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) were each assessed for severity by the investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement were assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. 0: 0% of BSA involvement with AD; 1: 1-9%; 2: 10-29%; 2: 30-49%; 4: 50-69%; 5: 70-89% and 6: 90-100% of BSA involvement with AD. Total score ranged from 0 (minimum) to 72 (maximum); higher scores indicated greater severity of AD. Participants who achieved EASI-75 were defined as participants with reduction of EASI score by ≥75% from baseline.
Percentage Of Participants With Reduction of Weekly Average of Daily Peak Pruritus Numerical Rating Scale (PP-NRS) of ≥4 Points From Baseline at Week 16 | Baseline (Day 1) and at Week 16
  The PP-NRS is a simple assessment tool that participants used to report the intensity of their pruritus (itch) during a daily recall period. Participants were asked to rate their worst itch on a 0 (no itch) to 10 (worst itch imaginable) NRS by answering the following question: For itch intensity, "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". The total score on the scale ranged from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicated worse symptoms. A minimum of 4 daily scores out of the 7 days is required to calculate the baseline average score.
Number of Participants With Weekly Average of Daily PP-NRS Reduction ≥4 From Baseline During The 16-Week Treatment Period | Baseline (Day 1) and Week 16
  The PP-NRS is a simple assessment tool that participants used to report the intensity of their pruritus (itch) during a daily recall period. Participants were asked to rate their worst itch on a 0 (no itch) to 10 (worst itch imaginable) NRS by answering the following question: For itch intensity, "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". The total score on the scale ranged from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicated worse symptoms. A minimum of 4 daily scores out of the 7 days is required to calculate the baseline average score.
Absolute Change From Baseline to Week 16 In EASI Score | Baseline (Day 1) to Week 16
  The EASI index is a validated investigator-administered scoring system used to measure the severity of clinical signs in AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) were each assessed for severity by the investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement were assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. 0: 0% of BSA involvement with AD; 1: 1-9%; 2: 10-29%; 2: 30-49%; 4: 50-69%; 5: 70-89% and 6: 90-100% of BSA involvement with AD. Total score ranged from 0 (minimum) to 72 (maximum); higher scores indicated greater severity of AD. Baseline was defined as the Day 1 assessment value.
Percentage of Participants Achieving EASI-50/90 (Reduction of EASI Score by ≥50% or ≥90% From Baseline) at Week 16 | Baseline (Day 1) and at Week 16
  The EASI index is a validated investigator-administered scoring system used to measure the severity of clinical signs in AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) were each assessed for severity by the investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement were assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. 0: 0% of BSA involvement with AD; 1: 1-9%; 2: 10-29%; 2: 30-49%; 4: 50-69%; 5: 70-89% and 6: 90-100% of BSA involvement with AD. Total score ranged from 0 (minimum) to 72 (maximum); higher scores indicated greater severity of AD. Participants who achieved EASI-50/90 were defined as participants with reduction of EASI score by ≥50% or ≥90% from baseline respectively.
Change From Baseline to Week 16 in Percent BSA of AD | Baseline (Day 1) to Week 16
  BSA affected by AD were assessed for each section of the body (the possible highest score for each region was: head and neck [10%], trunk including genitalia [30%], upper limbs [20%], lower limbs [40%]) and were reported as a percentage of all major body sections combined. Total score ranges from 0% to 100%. The higher score indicates a worse value and a lower score indicates a better value. Baseline was defined as the Day 1 assessment value.
Absolute Change From Baseline to Week 16 in Weekly Average of Daily PP-NRS | Baseline (Day 1) to Week 16
  The PP-NRS is a simple assessment tool that participants used to report the intensity of their pruritus (itch) during a daily recall period. Participants were asked to rate their worst itch on a 0 (no itch) to 10 (worst itch imaginable) NRS by answering the following question: For itch intensity, "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". The total score on the scale ranged from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicated worse symptoms. A minimum of 4 daily scores out of the 7 days is required to calculate the baseline average score. Baseline was defined as the Day 1 assessment value.
Percent Change From Baseline to Week 16 in Weekly Average of Daily PP-NRS | Baseline (Day 1) to Week 16
  The PP-NRS is a simple assessment tool that participants used to report the intensity of their pruritus (itch) during a daily recall period. Participants were asked to rate their worst itch on a 0 (no itch) to 10 (worst itch imaginable) NRS by answering the following question: For itch intensity, "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". The total score on the scale ranged from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicated worse symptoms. A minimum of 4 daily scores out of the 7 days is required to calculate the baseline average score. Baseline was defined as the Day 1 assessment value.
Percentage of Participants Achieving IGA*BSA-50/75/90 (Reduction of IGA*BSA by ≥50% or 75% or 90% From Baseline) At Week 16 | Baseline (Day 1) and at Week 16
  IGA is a static 5-point measure of disease severity based on an overall assessment of the skin lesions on a 5-point scale (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). Higher score indicated higher severity. Participants who achieved IGA*BSA-50-75-90 were defined as participants with reduction of IGA*BSA by ≥50% or 75% or 90% from baseline.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), Adverse Events of Special Interest (AESIs) and Study intervention Discontinuation | Baseline (Day 1) to 16 weeks
  An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were defined as AEs that developed, worsened or became serious during the treatment-emergent period. SAE was any AE that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. An AESI was an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the investigator to the Sponsor was required.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (9):
  - Antelope Valley Clinical Trials Site Number : 8400001, Northridge, California
  - Asthma and Allergy Associates, PC Site Number : 8400008, Colorado Springs, Colorado
  - Florida International Research Center Site Number : 8400002, Miami, Florida
  - Skin Sciences, PLLC Site Number : 8400005, Louisville, Kentucky
  - DS Research of Kentucky, LLC Site Number : 8400004, Louisville, Kentucky
  - Integrative Skin Care of MS/SKYCRNG Site Number : 8400011, Ridgeland, Mississippi
  - National Allergy and Asthma Research, LLC. Site Number : 8400007, North Charleston, South Carolina
  - Orion Clinical Research Site Number : 8400003, Austin, Texas
  - E.P.I.M.R.D dba Western Sky Research, Inc. Site Number : 8400009, El Paso, Texas
- Canada (7):
  - Investigational Site Number : 1240008, Red Deer, Alberta
  - Investigational Site Number : 1240013, Greater Sudbury, Ontario
  - Investigational Site Number : 1240001, London, Ontario
  - Investigational Site Number : 1240002, Markham, Ontario
  - Investigational Site Number : 1240011, Toronto, Ontario
  - Investigational Site Number : 1240007, Toronto, Ontario
  - Investigational Site Number : 1240004, Québec
- Chile (3):
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
- Czechia (4):
  - Investigational Site Number : 2030004, Olomouc
  - Investigational Site Number : 2030003, Pardubice
  - Investigational Site Number : 2030002, Pilsen
  - Investigational Site Number : 2030001, Prague
- Germany (2):
  - Investigational Site Number : 2760001, Bad Bentheim
  - Investigational Site Number : 2760002, Friedrichshafen
- Investigational Site Number : 5280001, Utrecht, Netherlands
- Poland (5):
  - Investigational Site Number : 6160001, Lodz, Lódzkie
  - Investigational Site Number : 6160005, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160008, Chojnice
  - Investigational Site Number : 6160002, Lodz
  - Investigational Site Number : 6160004, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT17207 Moderate-to-severe Atopic Dermatitis website — https://www.sanofistudies.com/eczema